CLINICAL TRIAL: NCT02474290
Title: Sorafenib for Prophylaxis of Leukemia Relapse in Allogeneic Hematopoietic Stem Cell Transplant Recipients With FLT3-ITD Positive Acute Myeloid Leukemia
Brief Title: Sorafenib for Prophylaxis of Leukemia Relapse in Allo-HSCT Recipients With FLT3-ITD Positive AML
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Peking University People's Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Zhujiang Hospital (Other); Xiangya Hospital of Central South University (Other); First People's Hospital of Chenzhou (Other); The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sorafenib-Flt3 AML-2015
Record Dates: First submitted 2015-06-14; First posted 2015-06-17 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2015-06

CONDITIONS: Acute Myeloid Leukemia; Hematopoietic Stem Cell Transplantation
Keywords: Acute Myeloid Leukemia; FLT3-ITD; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib group (Experimental): Sorafenib will be used from day 30 to 180 post-transplantation.
  Interventions: Drug: Sorafenib
- non-Sorafenib group (No Intervention)

INTERVENTIONS:
Drug: Sorafenib — The initial dose of sorafenib is 400 mg orally twice daily and is adjusted in case of suspected toxicity or resistance (dose range, 200-800 mg daily).
  Arms: Sorafenib group

SUMMARY:
The purpose of this study is to evaluate the efficacy of sorafenib for prophylaxis of leukemia relapse in allogeneic stem cell transplant (Allo-HSCT) recipients with FLT3-ITD positive acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
Internal tandem duplication of FMS-like tyrosine kinase 3 (FLT3-ITD) mutations have been reported in 20%-30% of patients with acute myeloid leukemia (AML). FLT3-ITD-positive AML patients have an inferior survival, primarily due to lower complete remission (CR) rate and higher relapse rate. Although allogeneic hematopoietic stem cell transplantation (allo-HSCT) improves the outcomes of some FLT3-ITD-positive AML, a significant number will suffer disease recurrence after allo-HSCT. Sorafenib, an inhibitor of multiple kinases including FLT3, has shown promising activity in FLT3-ITD-positive AML. Recent studies have shown that sorafenib monotherapy or in combination with chemotherapy are effective in attaining CR, but they do not have significant improvement in relapse. Currently, prophylactic use of sorafenib after allo-HSCT has been rarely reported, and whether it can improve outcomes of FLT3-ITD-positive AML remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* FLT3-ITD Positive AML
* Allo-HSCT Recipients

Exclusion Criteria:

* cardiac dysfunction (particularly congestive heart failure)
* hepatic abnormalities (bilirubin ≥ 3 mg/dL, aminotransferase> 2 times the upper limit of normal)
* renal dysfunction (creatinine clearance rate < 30 mL/min)
* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2015-06-20 (Actual); Primary Completion 2018-07-21 (Actual); Study Completion 2019-08-10 (Actual)

PRIMARY OUTCOMES:
Incidence of leukemia relapse | 1 year

SECONDARY OUTCOMES:
Overall survival | 3 year
leukemia-free survival | 3 year
Incidence of side effect of sorafenib | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Ravandi F, Cortes JE, Jones D, Faderl S, Garcia-Manero G, Konopleva MY, O'Brien S, Estrov Z, Borthakur G, Thomas D, Pierce SR, Brandt M, Byrd A, Bekele BN, Pratz K, Luthra R, Levis M, Andreeff M, Kantarjian HM. Phase I/II study of combination therapy with sorafenib, idarubicin, and cytarabine in younger patients with acute myeloid leukemia. J Clin Oncol. 2010 Apr 10;28(11):1856-62. doi: 10.1200/JCO.2009.25.4888. Epub 2010 Mar 8. PMID 20212254
- [Background] Metzelder SK, Schroeder T, Finck A, Scholl S, Fey M, Gotze K, Linn YC, Kroger M, Reiter A, Salih HR, Heinicke T, Stuhlmann R, Muller L, Giagounidis A, Meyer RG, Brugger W, Vohringer M, Dreger P, Mori M, Basara N, Schafer-Eckart K, Schultheis B, Baldus C, Neubauer A, Burchert A. High activity of sorafenib in FLT3-ITD-positive acute myeloid leukemia synergizes with allo-immune effects to induce sustained responses. Leukemia. 2012 Nov;26(11):2353-9. doi: 10.1038/leu.2012.105. Epub 2012 Apr 16. PMID 22504140
- [Derived] Xuan L, Wang Y, Yang K, Shao R, Huang F, Fan Z, Chi P, Xu Y, Xu N, Deng L, Li X, Liang X, Luo X, Shi P, Liu H, Wang Z, Jiang L, Lin R, Chen Y, Tu S, Zhang Y, Sun J, Huang X, Liu Q. Sorafenib maintenance after allogeneic haemopoietic stem-cell transplantation in patients with FLT3-ITD acute myeloid leukaemia: long-term follow-up of an open-label, multicentre, randomised, phase 3 trial. Lancet Haematol. 2023 Aug;10(8):e600-e611. doi: 10.1016/S2352-3026(23)00117-5. Epub 2023 Jul 3. PMID 37414062
- [Derived] Xu X, Fan Z, Wang Y, Huang F, Xu Y, Sun J, Xu N, Deng L, Li X, Liang X, Luo X, Shi P, Liu H, Chen Y, Tu S, Huang X, Liu Q, Xuan L. Effect of sorafenib maintenance on Epstein-Barr virus and cytomegalovirus infections in patients with FLT3-ITD AML undergoing allogeneic hematopoietic stem cell transplantation: a secondary analysis of a randomized clinical trial. BMC Med. 2022 Sep 2;20(1):282. doi: 10.1186/s12916-022-02479-x. PMID 36050712
- [Derived] Xuan L, Wang Y, Huang F, Fan Z, Xu Y, Sun J, Xu N, Deng L, Li X, Liang X, Luo X, Shi P, Liu H, Wang Z, Jiang L, Yu C, Zhou X, Lin R, Chen Y, Tu S, Huang X, Liu Q. Sorafenib maintenance in patients with FLT3-ITD acute myeloid leukaemia undergoing allogeneic haematopoietic stem-cell transplantation: an open-label, multicentre, randomised phase 3 trial. Lancet Oncol. 2020 Sep;21(9):1201-1212. doi: 10.1016/S1470-2045(20)30455-1. Epub 2020 Aug 10. PMID 32791048